CLINICAL TRIAL: NCT05292534
Title: Evaluation of the Clinical Benefit of the Hearing Aids Tinnitus Feature.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRF-481
Record Dates: First submitted 2022-03-09; First posted 2022-03-23 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-04

CONDITIONS: Hearing Loss, Sensorineural; Tinnitus
MeSH Terms: conditions — Hearing Loss, Sensorineural; Tinnitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Amplification-only (Active Comparator): Hearing aid will be fit to prescribed participant hearing loss.
  Interventions: Device: hearing aid amplification
- Amplification with added sound (Active Comparator): Hearing aid will be fit to prescribed participant hearing loss and an added sound will be activated on the hearing aid.
  Interventions: Device: hearing aid amplification with an added sound
- No intervention (No Intervention): Participants will return to their original unaided state.

INTERVENTIONS:
Device: hearing aid amplification — Hearing aid will be fit to prescribed participant hearing loss.
  Arms: Amplification-only
Device: hearing aid amplification with an added sound — Hearing aid will be fit to prescribed participant hearing loss and an added sound will be activated.
  Arms: Amplification with added sound

SUMMARY:
Participants with hearing loss and Tinnitus will wear hearing aids with amplification-only or with an added sound, and have their tinnitus level evaluated before and after intervention.

DETAILED DESCRIPTION:
2 groups of adults with hearing loss and chronic bothersome tinnitus and no experience with amplification will participate in a cross over intervention study with 2 conditions of 4 weeks each: 1. fit with hearing aid (HA) amplification-only, and 2. fit with HA amplification with an added sound, returning to their original unaided condition after undergoing the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss
* candidate for hearing aid amplification
* Bothersome chronic tinnitus (3 months+)

Exclusion Criteria:

* age less than 18 years
* normal hearing
* tinnitus presence for less than 3 months
* tinnitus not bothersome enough to warrant intervention
* non hearing aid candidates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Sun, Ph.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- The State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Henry JA, Griest S, Thielman E, McMillan G, Kaelin C, Carlson KF. Tinnitus Functional Index: Development, validation, outcomes research, and clinical application. Hear Res. 2016 Apr;334:58-64. doi: 10.1016/j.heares.2015.06.004. Epub 2015 Jun 12. PMID 26074306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 participants signed the consent form and met study criteria
Pre-assignment Details: 38 participants were randomly assigned into one of two groups. Out of the 38 participants, 8 dropped out during the study. There were 2 study groups in this cross-over study, and final numbers were 15 participants in each group.
Groups:
- Amplification-only, Then Amplification With an Added Sound, Then Intervention Withdrawal: 3 study conditions (4 weeks each):
  1. Hearing aid amplification-only,
  2. Hearing aid amplification with an added sound,
  3. intervention withdrawal.
  Hearing aid was fit to prescribed participant hearing loss for 4 weeks during the 1st intervention period.
  Then the participants wore the same study hearing aids for another 4 weeks with an added sound to the amplification setting.
  Then the participants returned the hearing devices to the investigator and were re-assessed 4 weeks after intervention withdrawal.
- Amplification With Added Sound, Then Amplification-only, Then Intervention Withdrawal: 3 study conditions (4 weeks each):
  1. Hearing aid amplification with an added sound,
  2. Hearing aid amplification-only,
  3. intervention withdrawal.
  Hearing aid was fit to prescribed participant hearing loss and an added sound activated on the hearing aid and worn for 4 weeks during the 1st intervention period.
  Then the participants wore the same study hearing aids for another 4 weeks without the added sound to the amplification setting.
  Then the participants returned the hearing devices to the investigator and were re-assessed 4 weeks after intervention withdrawal.
Period: Overall Study
Arm/Group | Amplification-only, Then Amplification With an Added Sound, Then Intervention Withdrawal | Amplification With Added Sound, Then Amplification-only, Then Intervention Withdrawal
Started | 18 (First participant seen on Jun3 2022) | 20
Completed | 15 | 15
Not Completed | 3 | 5
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Group 1 and Group 2 had 15 participants/each.
Groups:
- Cross Over Design, 2 Groups of Participants: First Group: started with amplification-only as a 1st intervention, and switched to amplification+noiser Second Group: started with amplification+noiser as a 1st intervention, and switched to amplification-only
Arm/Group | Cross Over Design, 2 Groups of Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Table above present the mean age (and standard deviation) of each separate group of 15 participants.
  years
    Group 1: number analyzed (Participants) | 15
    Group 1 | 62.2 (9.5)
    Group 2: number analyzed (Participants) | 15
    Group 2 | 60.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 30 participants divided into 2 groups of 15 participants/each.
  Participants
    Group 1: number analyzed (Participants) | 15
    Group 1: Female | 8
    Group 1: Male | 7
    Group 2: number analyzed (Participants) | 15
    Group 2: Female | 4
    Group 2: Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
TFI [Mean (Standard Deviation); unit: points] — Population: 15 participants in each of the 2 groups, totaling 30 participants in the study.
  points
    Group 1: number analyzed (Participants) | 15
    Group 1 | 50 (16.1)
    Group 2: number analyzed (Participants) | 15
    Group 2 | 36.2 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index Evaluation (TFI)
Description: Tinnitus Functional Index (TFI) questionnaire results, ranging from 0 to 100, with higher numbers indicating more severe (worse) Tinnitus interference in the person's quality of life.
Time Frame: TFI collected before intervention to serve as a baseline. TFI change from baseline will be assessed after each study condition, which will last 4 weeks/each.
Population: Repeated measures. Participants served as their own control.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amplification-only | Amplification With Added Sound | No Intervention
Number analyzed (Participants) | 30 | 30 | 30
units on a scale
  Group 1: number analyzed (Participants) | 15 | 15 | 15
  Group 1 | 35.6 (20) | 32 (21.9) | 44.8 (22.2)
  Group 2: number analyzed (Participants) | 15 | 15 | 15
  Group 2 | 36.2 (19.0) | 34.4 (19.7) | 40.4 (16.5)

ADVERSE EVENTS:
Time Frame: 10 months (Between Nov 2022 until September 2023).
Description: Safety population included all participants in this study, who experienced at least one intervention mode.
Arm/Group | Amplification-only | Amplification With Added Sound | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amplification-only (N=30) | Amplification With Added Sound (N=30) | No Intervention (N=30)
Acquired COVID (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infection after swimming (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Body ache after general incidents happening during the trial period (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) — Events were: body ache after moving furniture, body ache after falling in the bathroom at night, mouth discomfort after being stuck open at the dentist during a procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT05292534/Prot_SAP_000.pdf